CLINICAL TRIAL: NCT05844007
Title: A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana
Brief Title: A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana Year 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Lauren Davis, Assistant Professor, Montana State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MontanaSUYear4; 5P20GM104417 (NIH)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Trauma and Stressor Related Disorders
MeSH Terms: conditions — Trauma and Stressor Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High School Students: Remote Delivery (Experimental): Remote delivery of trauma-informed yoga session for high school students
  Interventions: Behavioral: Trauma-Informed Yoga
- High School Students: Face-to-Face Delivery (Experimental): Face-to-face delivery of trauma-informed yoga session for high school students
  Interventions: Behavioral: Trauma-Informed Yoga
- Teachers: Remote Delivery (Experimental): Remote delivery of trauma-informed yoga session for teachers
  Interventions: Behavioral: Trauma-Informed Yoga

INTERVENTIONS:
Behavioral: Trauma-Informed Yoga — Trauma-informed yoga intervention, delivered either in-person or remotely for 6 weeks, twice weekly for 45 minutes sessions

SUMMARY:
Compared to U.S. urban counterparts, rural residents face major barriers to using health care services. Challenges include shortages of services, long distances to existing services, and stigma regarding mental illness in isolated communities. These difficulties hold true for Montana, but especially for adolescents. The objective of A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana is to improve stress-related mental and physical health outcomes for adolescents and educators in rural Montana through school-based, trauma-informed yoga exercises. This project builds on investigators' previous research (including a two-year CAIRHE pilot study, 2019-21) to promote positive youth development by simultaneously intervening with students and teachers with a trauma-informed yoga intervention. Geographic isolation and resulting lack of resources for many Montanan schools indicates a need for novel, school-centered interventions to address the needs of rural adolescents; yoga can benefit youth and teacher wellbeing.

DETAILED DESCRIPTION:
In Year 2, investigators will expand the study to pilot test a remote delivery for students and teachers in rural schools through virtual delivery (in addition to an in-person high school student intervention at the school district of Aim 1. Primary outcomes for teachers will assess career satisfaction/self-efficacy; primary outcomes for students will assess depression/anxiety symptomology. Effects on secondary mental/physical health outcomes will be drawn from survey results, cortisol levels, and heart rate variability measures (collected pre/post).

Investigators will then determine which intervention design was more effective with students (in-person vs. remote) between the two years of this feasibility study through an outcome evaluation. Comparisons of mental and physical health outcomes will be examined by the research team using cohort data drawn from participants' physiological data and survey results.

The short-term public health impact of this study is to improve the mental and physical health of rural Montana youth and teachers through a novel, school-based intervention. If successful, this study's long-term public health impact will reduce rates of anxiety and depression and improve physical health in geographically isolated settings.

ELIGIBILITY:
Inclusion Criteria:

* Any teacher currently employed by the Livingston or Gardiner school district who wishes to participate in the intervention (up to 45 participants)
* Any freshmen student enrolled in pre-selected PE classes at Park High School in Livingston Montana
* Any PE student enrolled in pre-selected PE classes at Gardiner High School in Gardiner Montana

Exclusion Criteria:

* Any students that are not enrolled in pre-selected PE classes at Park or Gardiner High Schools in Southwest Montana

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Adams, MD, Ph.D, Study Director — Montana State University
Locations (1):
- Park High School, Livingston, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
Started | 22 | 18 | 43
Completed | 22 | 18 | 43
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery | Total
Number analyzed (Participants) | 22 | 18 | 43 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 18 | 0 | 40
  Between 18 and 65 years | 0 | 0 | 42 | 42
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 37 | 57
  Male | 11 | 9 | 6 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cortisol Levels [Mean (Standard Deviation); unit: micrograms per deciliter] | 0.3 (.40) | .43 (.38) | .16 (.11) | 0.3 (.3)

OUTCOME MEASURES:

1. Primary Outcome: Salivary Cortisol Levels
Description: Participants will provide a saliva sample in which cortisol levels will be analyzed through salivary assay kits (through Salimetrics.com). Samples will be collected on the first day of the intervention (week 1) and on the last day of the intervention (week 6) to determine if the intervention has improved stress levels (as indicated by a reduction in cortisol levels). A biostatistician will provide analysis and conclusion of these samples at the conclusion of the study
Time Frame: Pre-Intervention, first day of Week 1 and post-intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: micrograms per deciliter
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
Number analyzed (Participants) | 22 | 18 | 43
micrograms per deciliter
  Post-Intervention: Last day of week 6 | .33 (.2) | .25 (.13) | .15 (.11)
  Pre-Intervention: First day of week 1 | .30 (.40) | .43 (.38) | .16 (.11)

2. Primary Outcome: Patient Health Questionnaire
Description: This 9 item questionnaire is designed to evaluate severity of depressive symptoms in participants. It is scored on a Likert scale from 0 (not at all) to 3 (nearly every day) on items linked to depression indicators. The minimum score is a 0 and the maximum score is a 27, and a reduction in score from pre- to post-assessment indicates an improvement in symptomology.
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
Number analyzed (Participants) | 22 | 18 | 43
score on a scale
  Pre-Intervention: First day of Week 1 | 11.84 (7.02) | 6.47 (4.60) | 7.1 (4.8)
  Post-Intervention, last day of Week 6 | 8.67 (5.86) | 4.92 (4.69) | 4.5 (3.6)

3. Primary Outcome: Generalized Anxiety Disorder-7 Anxiety Scale
Description: This 7 item questionnaire is based on a likert scale of 0 (not at all) to 3 (nearly every day) for items related to anxiety disorders. The lowest score is a zero and the maximum score is a 21. A reduction in score from pre- to post-assessment indicates an improvement in symptomology.
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
Number analyzed (Participants) | 22 | 18 | 43
score on a scale
  Pre-Intervention: First day of Week 1 | 9.45 (5.62) | 7.84 (5.36) | 7.9 (5.1)
  Post-Intervention, last day of Week 6 | 8.22 (4.57) | 6.06 (5.02) | 5.4 (4.4)

4. Primary Outcome: Heart Rate Variability
Description: Participants enrolled will have their heart rate data measured by the Biopac BioNomadix PPG & EDA System with Pulse Transduce to determine heart rate variability. Due to circumstances beyond the research team's control, only teachers at one study site were able to provide heart rate variability data, so fewer than our total enrollment was able to provide this data.
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
Number analyzed (Participants) | 21 | 14 | 29
beats per minute (bpm)
  Pre-Intervention: First day of Week 1 | 72.55 (13.27) | 70.29 (10.28) | 68.46 (11.00)
  Post-Intervention, last day of Week 6 | 73.34 (11.73) | 69.00 (8.85) | 70.87 (12.41)

5. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: The CD-RISC 10 is a unidimensional self-reported scale consisting of 10-items measuring resilience. Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4. The minimum score possible is a 0 and the maximum score is a 40. A higher score indicates an improvement (increased resilience).
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
Number analyzed (Participants) | 22 | 18 | 43
score on a scale
  Pre-Intervention: First day of Week 1 | 26.64 (8.17) | 25.68 (6.52) | 28.8 (4.9)
  Post-Intervention, last day of Week 6 | 25.56 (7.76) | 27.33 (6.06) | 29.2 (4.3)

6. Secondary Outcome: Professional Quality of Life Index (Pro-QOL)
Description: Teachers will complete this self-reporting scale consisting of 30 items measuring levels of compassion satisfaction, secondary trauma, and professional burnout. Respondents rate items on a 5 point Likert scale ranging from 0 (never) to 5 (very often). Scores within each subscale were added together to produce a mean for each subscale; subscale means were then averaged together for a total mean score. The minimum score for each subscale is a 0, and the maximum score for each subscale is a 50. Reduced scores indicate an improvement in burnout and secondary trauma.
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teachers: Remote Delivery
Number analyzed (Participants) | 43
score on a scale
  Pre-Intervention: First day of Week 1 | 32.6 (5.27)
  Post-Intervention, last day of Week 6 | 31.27 (5.07)

7. Secondary Outcome: Teachers' Sense of Self-Efficacy (Short Form)
Description: Teachers will complete this self-reporting scale consisting of 12 items measuring levels of self-perceived levels of impact on student engagement, instructional strategies, and classroom management. Respondents rate items on a 9 point Likert scale ranging from 0 (nothing) to 9 (a great deal). The minimum score possible is a 0 and the maximum score is a 90. Subscale scores were averaged together to produce a single mean. Higher mean scores indicate improvements in self-perceptions of self-efficacy.
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teachers: Remote Delivery
Number analyzed (Participants) | 43
score on a scale
  Pre-Intervention: First day of Week 1 | 83.2 (11.8)
  Post-Intervention, last day of Week 6 | 81.5 (12.4)

8. Secondary Outcome: PROMIS Sleep Disturbance Scales
Description: Participants will complete this self-reporting scale consisting of 8 items measuring perceived levels of sleep quality over the previous 7 days. Items are scored on a Likert scale ranging from 1 (not at all) to 5 (very much). The minimum score possible is 8 and the maximum score is a 40. Lower scores indicate an improvement in sleep quality, and higher scores indicate increased severity of sleep disturbances.
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
Number analyzed (Participants) | 22 | 18 | 43
score on a scale
  Pre-Intervention: First day of Week 1 | 22.27 (2.80) | 23.00 (3.18) | 22.1 (2.9)
  Post-Intervention, last day of Week 6 | 23.39 (3.45) | 22.28 (2.47) | 21.2 (2.9)

9. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: Teachers will complete this self-reporting scale consisting of 20 items measuring traumatic stress symptoms in the previous month. Items are scored on a Likert scale from 0 (not at all) to 4 (extremely). The minimum score possible is a 0 and the maximum score is an 80. Lower scores indicate improvements in traumatic stress symptoms, and higher scores worsening levels of traumatic stress in respondents.
Time Frame: Pre-Intervention: First day of Week 1 and Post-Intervention, last day of Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teachers: Remote Delivery
Number analyzed (Participants) | 43
score on a scale
  Pre-Intervention: First day of Week 1 | 19.5 (12.9)
  Post-Intervention, last day of Week 6 | 12.8 (10)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | High School Students: Remote Delivery | High School Students: Face-to-Face Delivery | Teachers: Remote Delivery
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/43
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT05844007/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT05844007/ICF_001.pdf